CLINICAL TRIAL: NCT05020561
Title: Adjustment to Life After Breast Cancer Treatment: Can a Life-Coach Make a Difference
Brief Title: Life After Breast Cancer - Impact of a Life Coach
Acronym: Lifecoach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Quebec Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Dr. Sarkis Meterissian, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-7735
Record Dates: First submitted 2021-08-12; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Survivorship; Breast Cancer
Keywords: Breast Cancer Survivorship; Post-traumatic Growth; Quality of Life; Fear of Recurrence; Randomized controlled trial
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - Group and Individual (Experimental): Participants in this experimental Arm 1 will receive the 3 group sessions followed by 4 to 5 individual coaching sessions via phone calls that last 60 minutes each.
  Interventions: Behavioral: Group life-coaching; Behavioral: Individual life-coaching
- Arm 2 - Group only (Experimental): Arm 2 will receive only the first 3 Life coach sessions (group session).
  Interventions: Behavioral: Group life-coaching
- Arm 3 - Routine care (No Intervention): Arm 3 will receive routine care by the Breast clinic team for the entire course of the study.

INTERVENTIONS:
Behavioral: Group life-coaching — Group coaching sessions will be focusing on providing material and tools that guide the participants in the transition from cancer treatment to survivorship. All activities of the group session will be following the "After Cancer Passport" document.
  Arms: Arm 1 - Group and Individual; Arm 2 - Group only
Behavioral: Individual life-coaching — In the individual coaching sessions, the life-coach will provide guidances that help the participants to put tools into actions. All activities are outlined in the After Cancer Passport. Participants will use their Passport for each individual coaching session to outline their objectives and indicators of success. The life coach will also assign activities, such as self-reflection, for the participants to complete between each session.
  Arms: Arm 1 - Group and Individual

SUMMARY:
The objectives of our intervention are to

1. Ease the transition between cancer treatment and active life, and
2. Allow breast cancer survivors to take control of their lives.

The primary objective of this study is to:

1) Determine whether individual life coaching (i.e., individualized guidance that helps to put resources into action) can significantly improve quality of life and post-traumatic growth among women who have been recently treated with breast cancer.

It is hypothesized that:

1. Participants who receive both "group coaching sessions" and "individualized coaching sessions" will report greater post-traumatic growth and quality of life, and less fear of cancer recurrence when compared to the breast cancer survivors who received only the group coaching sessions or usual care.
2. Participants who receive only the group coaching sessions will report greater post-traumatic growth and quality of life, and lesser fear of cancer recurrence when compared to the participants who receive usual care.

ELIGIBILITY:
Inclusion Criteria:

1. have been diagnosed with stage I, II, or III breast cancer;
2. are female breast cancer patients over the age of 18;
3. have completed anti-cancer treatment via surgery and/or chemotherapy and /or radiation therapy at the McGill University Health Centre Breast Clinic;
4. are fluent in written and spoken English or French;
5. are alert and oriented and capable of giving informed consent;
6. have an Internet connection at home that supports participation in coaching sessions via videoconferencing (zoom).

Exclusion Criteria:

1. have a recurrence of breast cancer;
2. are diagnosed with a second cancer;
3. are diagnosed with stage IV breast cancer due to their worse prognosis; and 4) have an active psychiatric diagnosis that would render adherence to the study problematic.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Post-traumatic growth (PTG) assessed by the Post-Traumatic Growth Inventory (PTGI) | 12 months
  The PTGI consists of 21 items, the response scale is a 6-point Likert scale asking respondents the degree to which changes occurred in their lives as a result of the crisis, where 0 represented "I did not experience this change" and 5 represented "I experienced this change to a very great degree". The PTGI is composed of 5 subscales, with 5 items measuring the construct New Possibilities, 7 items measuring the construct Relating to Others, 4 items measuring the construct Personal Strength, 3 items measuring the construct Appreciation of Life and 2 items measuring the construct Spiritual Change. The scores are summed to provide an overall measure of post-traumatic growth ranging from 0 - 105 where higher scores indicate more reported growth.

SECONDARY OUTCOMES:
Change from baseline Fear of cancer recurrence (FCR) assessed by the Cancer Worry Scale (CWS) | 12 months
  The CWS is a six-item scale designed to measure worry about the risk of developing cancer and the impact of worry on daily functioning. The six items are rated on a 4-point Likert scale ranging from 1 ("never") to 4 ("almost always"). Possible scores range from 6 to 24 with higher scores indicating more worry.
Change from baseline Quality of life (QoL) assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS)-Preference | 12 months
  The PROPr is a 31-item instrument assessing eight domains (29 items) (i.e., anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, ability to participate in social roles and activities, and pain intensity), and Cognitive Function Abilities (2 items). Raw scores generated for each domain are transformed into T scores; higher PROMIS T scores indicate greater endorsement of the construct being assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Cedar's Breast Clinic, Royal Victoria Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: will be submitted to the International Journal of Clinical Trials (IJCT) in November 2022

REFERENCES:
- [Derived] Tock WL, Maheu C, Blondin S, Lee V, Neuman S, Meterissian S. The Effect of Life Coaching on Post-Traumatic Growth and Well-Being in Breast Cancer Survivors: A Randomized Controlled Trial. Psychooncology. 2025 Oct;34(10):e70295. doi: 10.1002/pon.70295. PMID 41068064